CLINICAL TRIAL: NCT02692547
Title: Feasibility Study to Evaluate the Hybrid-Logic Closed Loop System in Type 1 Diabetes
Acronym: DREAMED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Cancelled
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP312
Record Dates: First submitted 2015-12-03; First posted 2016-02-26 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hybrid-logic closed loop system (Other): All patients get to wear the pump. only 1 arm. There is no comparator in this study, as all patients wear the pump.
  Interventions: Device: Hybrid-logic closed loop system

INTERVENTIONS:
Device: Hybrid-logic closed loop system — All patients get to wear the pump

SUMMARY:
The purpose of this study is to collect data on the feasibility of the HLCL system in a camp setting.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, in clinic Investigation in subjects with type 1 diabetes on insulin pump therapy.

Run-in Period A total of up 10 subjects will be enrolled (age 18-25). A minimum of 6 days run-in period with the 640G (sensor augmented pump) will be used to collect sensors and insulin data and to allow the subject to become familiar.

Study Period - Camp Following the run-in period subjects will participate in a 5 day, 4 night study period in an camp setting during which the CL feature will be studied.

Subjects will receive 3 meals each day, one night they receive a high fat dinner, one morning they will receive breakfast high in carbohydrates.

Subjects will be asked to exercise for up to 60 minutes on one day during their study period.

Subjects will be asked to take a minimum of 5 fingersticks a day (before each meal, morning and before bedtime)

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes duration > 1 year since diagnosis
2. Sensor augmented Pump for at least 6 months
3. Age 18-25
4. A1C <10.0 at time of screening visit
5. Willing to follow study instructions
6. Willing to perform ≥ 5 finger stick blood glucose measurements daily
7. Willing to perform required sensor calibrations
8. Patient capable of reading and understand instructions in English

Exclusion Criteria:

1. Subject is unable to tolerate tape adhesive in the area of sensor placement
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject has a positive pregnancy screening test
5. Subject is female, sexually active without the use of contraception, and plans/able to become pregnant during the course of the study and is not using an acceptable method of contraception
6. Subject has had a hypoglycemic seizure within the past 6 months prior to screening visit
7. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit
8. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit
9. Subject has a history of a seizure disorder
10. Subject has central nervous system or cardiac disorder resulting in syncope
11. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
12. Subjects with hematocrit lower than the normal reference range per POC or local lab testing
13. Subjects with a history or findings on screening electrocardiogram (EKG) of any cardiac arrhythmia, including atrial arrhythmias
14. Subjects with a history of adrenal insufficiency
15. Subjects with history of migraines that have occurred at least 2 times in the last 3 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Descriptive endpoints | after 4 days of camp
  Time in different range SG 70 mg/dL ≤ SG ≤ 180 mg/dL

SECONDARY OUTCOMES:
Descriptive endpoints | after 4 days of camp
  Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Philip, MD, Principal Investigator — National Center for Childhood Diabetes, Schneider Children's Medical Center of Israel

IPD SHARING:
Plan to Share IPD: No